CLINICAL TRIAL: NCT07261345
Title: The Safety and Efficacy of Allogenic Anti-CD19/BCMA CAR-T Cell Therapy for Refractory Graves' Disease
Brief Title: Allogeneic Anti-CD19/BCMA CAR-T for Refractory Graves' Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-711
Record Dates: First submitted 2025-11-23; First posted 2025-12-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Graves' Disease
Keywords: CAR-T; TSH receptor antibody; refractory Graves' disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will receive a single dose of allogenic anti-CD19/BCMA CAR-T (RD06-05).
  Interventions: Biological: allogenic anti-CD19/BCMA CAR-T

INTERVENTIONS:
Biological: allogenic anti-CD19/BCMA CAR-T — Participants will receive a single infusion of allogenic anti-CD19/BCMA CAR-T (RD06-05).

SUMMARY:
Graves' disease is an autoimmune thyroid disorder in which autoantibodies against the thyroid-stimulating hormone receptor (TRAb) lead to excessive thyroid hormone production and systemic complications, as well as thyroid eye disease and pretibial myxedema in some cases. Patients with refractory Graves' disease often fail to achieve durable remission despite prolonged antithyroid medication.

This study aims to evaluate the safety and efficacy of RD06-05, an allogeneic dual CD19/BCMA CAR-T therapy, in participants with refractory Graves' disease, and will provide preliminary evidence on whether dual-targeting CAR-T therapy can induce sustained remission of refractory Graves' disease.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following inclusion criteria to be eligible for this study):

* Refractory Graves' disease, defined as meeting at least one of the following: a) Continuous treatment with antithyroid drugs (ATDs) for ≥3 years without achieving criteria for drug discontinuation. b) Meeting criteria for drug discontinuation but experiencing ≥2 relapses after withdrawal.
* Positive serum TRAb.
* Willing to voluntarily participate in this clinical study, able to sign informed consent, and compliant with follow-up requirements.

Exclusion Criteria (Participants will be excluded if any of the following conditions apply):

* History of severe drug allergies or allergic constitution.
* Presence or suspected presence of uncontrolled or active infections (including bacterial, fungal, viral, or other pathogens) requiring systemic or intravenous treatment.
* Presence of central nervous system disorders (including epilepsy, psychosis, cerebrovascular accident, encephalitis, CNS vasculitis, etc).
* Presence of clinically significant heart diseases (e.g., angina pectoris, myocardial infarction, heart failure, severe arrhythmias, etc).
* Subjects with congenital immunoglobulin deficiency.
* Subjects with malignancy (current or past), except for conditions deemed cured and with no risk of recurrence based on investigator assessment.
* Positive viral serology, including any of the following: Hepatitis B surface antigen (HBsAg)-positive, or hepatitis B core antibody (HBcAb)-positive with HBV DNA above the upper limit; Hepatitis C virus (HCV) antibody-positive with detectable HCV RNA; Human immunodeficiency virus (HIV) antibody-positive; Positive syphilis test.
* Severe psychiatric disorder or significant cognitive impairment that may affect compliance.
* Hematologic dysfunction, including: a) White blood cell count < 3.5 × 10⁹/L; b) Neutrophil count < 1.8 × 10⁹/L; c) Hemoglobin < 110 g/L.
* Hepatic dysfunction, defined as any of the following: Alanine aminotransferase (ALT) > 3 × ULN; Aspartate aminotransferase (AST) > 3 × ULN; Total bilirubin (TBIL) > 2.5 × ULN.
* Renal dysfunction: creatinine clearance rate (CrCl) < 60 mL/min (Cockcroft-Gault formula).
* Left ventricular ejection fraction (LVEF) < 55%.
* Coagulation abnormalities, defined as either: International normalized ratio (INR) > 1.5 × ULN; Prothrombin time (PT) > 1.5 × ULN.
* Participation in another clinical trial within 3 months prior to enrollment.
* Pregnant or breastfeeding women, or women planning to become pregnant.
* Any other condition that, in the opinion of the investigator, would make the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (AEs) | From baseline to 12 months after infusion of CAR-T cells
Remission of Graves' disease | From baseline to 12 months after infusion of CAR-T cells
  Proportion of remission will be calculated throughout 12 months after infusion of CAR-T cells. Remission is defined as euthyroid status without anti-thyroid medication.

SECONDARY OUTCOMES:
Proportion of participants with ≥50% reduction of anti-thyrotropin receptor antibody (TRAb) | From baseline to 12 months after infusion of CAR-T cells
  Percentage of participants achieving a ≥50% reduction of TRAb throughout 12 months after infusion of CAR-T, as compared with baseline.
Proportion of participants with ≥50% reduction of thyroid stimulating immunoglobulin (TSI) | From baseline to 12 months after infusion of CAR-T cells
  Percentage of participants achieving a ≥50% reduction of TSI throughout 12 months after infusion of CAR-T, as compared with baseline.
Change of TRAb levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  TRAb levels will be measured from baseline to 12 months after infusion of CAR-T cells
Change of TSI levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  TSI levels will be measured from baseline to 12 months after infusion of CAR-T cells
Change of thyroid gland volume compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  Size of the thyroid will be measured and calculated by ultrasound from baseline to 12 months after infusion of CAR-T cells
Change of thyroid peroxidase antibody (TPOAb) levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  TPOAb levels will be measured from baseline to 12 months after infusion of CAR-T cells
Change of thyroglobulin antibody (TgAb) levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  TgAb levels will be measured from baseline to 12 months after infusion of CAR-T cells.
Change of serum free T3 (FT3) levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  FT3 levels will be measured from baseline to 12 months after infusion of CAR-T cells
Change of serum free T4 (FT4) levels compared to baseline | From baseline to 12 months after infusion of CAR-T cells
  FT4 levels will be measured from baseline to 12 months after infusion of CAR-T cells
Cmax of CAR-T cells after infusion | Day 0 to Day 28
  Peak peripheral blood concentration of CAR-T cells (RD06-05 ) following infusion, measured by flow cytometry.
Tmax of CAR-T cells after infusion | Day 0 to Day 28
  Time to reach maximum observed concentration (Tmax) of CAR-T cells (RD06-05).
Dynamic change of circulating CAR-T cell count | From baseline to 3 months after infusion
Dynamic change of CAR transgene copy number | From baseline to 3 months after infusion
Dynamic change of peripheral B lymphocyte cell counts | From baseline to 12 months after infusion of CAR-T cells.
Dynamic change of serum interleukin-6 | From baseline to 3 months after infusion of CAR-T cells.
Dynamic change of serum tumor necrosis factor α (TNF-α) | From baseline to 3 months after infusion of CAR-T cells.
Dynamic change of serum immunoglobulin levels | From baseline to 12 months after infusion

OTHER OUTCOMES:
BCR repertoire dynamics (Exploratory) | From baseline to 12 months after infusion
  High-throughput sequencing of B-cell receptor (BCR) repertoires
TCR repertoire dynamics (Exploratory) | From baseline to 12 months after infusion
  High-throughput sequencing of T-cell receptor (TCR) repertoires

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After publication.
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).